CLINICAL TRIAL: NCT05833880
Title: Use of Complementary and Alternative Medicine in Children and Adults With Atopic Dermatitis: a Single-center Prospective Observational Study
Brief Title: Use of Complementary and Alternative Medicine in Children and Adults With Atopic Dermatitis
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Anne Claire BURSZTEJN, Director, Head of Dermatology, Principal Investigator, Clinical Professor, Central Hospital, Nancy, France
Other Study IDs: 2023-A00605-40
Record Dates: First submitted 2023-04-02; First posted 2023-04-27 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; Atopic Eczema; Complementary and Alternative Medicine
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Atopic dermatitis patients
  Interventions: Behavioral: Self-administered questionnaire

INTERVENTIONS:
Behavioral: Self-administered questionnaire — Self-administered questionnaire regarding complementary and alternative medicine use

SUMMARY:
Complementary and alternative medicine are increasingly used all around the world and more specifically in chronic diseases such as atopic dermatitis. Sociodemographic and disease determinants associated with their use remain unclear. Moreover, most of studies involved children and little data are available for adults.

The main objective of this study is to identify factors associated with complementary and alternative medicine use in children and adults suffering from atopic dermatitis. The secondary objectives are to determine the prevalence of complementary and alternative medicine use, the main forms used and their modalities of use, patients' motivations for using these therapies and sources of information.

Patients of all ages consulting for their atopic dermatitis at the dermatology or pediatric allergology department of Nancy University Hospital over a 6 months period will be asked to fill out a questionnaire about their pathology and their use of complementary and alternative medicine. This questionnaire will be collected before they leave the hospital.

ELIGIBILITY:
Inclusion Criteria:

* All patients, adults or children, without age limit;
* Patients visiting the dermatology or pediatric allergology department of Nancy University Hospital;
* Patients with atopic dermatitis confirmed on clinical examination by the physician;
* Patients with a history of atopic dermatitis or newly diagnosed patients;
* Patient affiliated to a social security plan or beneficiary of such a plan;
* Patients who understand French and are able to complete a self-administered questionnaire or have the option of assistance in completing it.

Exclusion Criteria:

* Patient with at least one other dermatological pathology or non-atopic eczema (contact eczema, ...);
* Patient without a confirmed diagnosis of atopic dermatitis by a physician;
* Patient who has already completed the questionnaire during a previous consultation;
* Pregnant and breastfeeding women;
* Refusal of the patient or at least one of the parents for children;
* Patient placed under court protection, guardianship or curatorship;
* Patient deprived of liberty by a judicial or administrative decision.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients of all ages suffering from atopic dermatitis visiting the dermatology or pediatric allergology department of Nancy University Hospital
Sampling Method: Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2023-08-03 (Actual); Study Completion 2023-08-03 (Actual)

PRIMARY OUTCOMES:
Binary variable: use of complementary and alternative medicine (yes/no) | Baseline (J0)
  Binary variable: use of complementary and alternative medicine (yes/no), variable collected by questionnaire, as reported by the patient (or the patient's parents)

SECONDARY OUTCOMES:
Percentage of patients using complementary and alternative medicine in relation to the total number of patients included in the study | Baseline (J0)
  Percentage of patients using complementary and alternative medicine in relation to the total number of patients included in the study, variable collected by questionnaire according to the patient's declaration (use or not use of complementary and alternative medicine) and then calculated
Forms of complementary and alternative medicine used | Baseline (J0)
  Forms of complementary and alternative medicine used, variable collected by questionnaire, as reported by the patient (or the patient's parents)
Modalities of use of complementary and alternative medicine | Baseline (J0)
  Modalities of use of complementary and alternative medicine, variable collected by questionnaire, as reported by the patient (or the patient's parents)
Patients' motivations for using complementary and alternative medicine | Baseline (J0)
  Patients' motivations for using complementary and alternative medicine, variable collected by questionnaire, as reported by the patient (or the patient's parents)
Sources of information regarding complementary and alternative medicine | Baseline (J0)
  Sources of information regarding complementary and alternative medicine, variable collected by questionnaire, as reported by the patient (or the patient's parents)

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Claire Bursztejn, Principal Investigator — University Hospital of Nancy, France
Locations (1):
- University Hospital of Nancy, Nancy, France